CLINICAL TRIAL: NCT03001609
Title: An Open-Label, Non-Randomized, Single-Center Study to Determine the Absorption, Metabolism and Excretion of A Single Dose [14C] AC0010 in Patients With Advanced NSCLC
Brief Title: Study to Investigate the Absorption, Metabolism and Excretion of [14C] AC0010 in Patients With Advanced NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou ACEA Pharmaceutical Research Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC201606AVTN06
Record Dates: First submitted 2016-12-19; First posted 2016-12-23 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — abivertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AC0010 (Experimental): each participant will be given a single dose of 14C-labeled AC0010
  Interventions: Drug: AC0010

INTERVENTIONS:
Drug: AC0010 — Oral dose of 14C-labeled AC0010 suspension including 200 mg/83μCi[14C]
  Other Names: 14C-labeled AC0010 oral; AC0010MA

SUMMARY:
The purpose of this study is to investigate Pharmacokinetics parameters of a single dose [14C] AC0010 in male Patients With Advanced NSCLC.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the Absorption, Metabolism, Excretion and Pharmacokinetics of a single dose [14C] AC0010 in male Patients With Advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* signed and dated informed consent
* histologically or cytologically confirmed diagnosis of local advanced or recurrent NSCLC
* failed to the treatment of EGFR-TKI and harbored T790M mutation
* male, Age 18~ 65, have a body mass index (BMI) >19 kg/m2
* ECOG PS:0-1,Life expectancy of more than 3 months
* main organs function is normal, laboratory values as listed below: blood test without blood transfusion within 14 days

  1. Haemoglobin >100 g/L
  2. Absolute neutrophil count ≥2.0x10^9/L or WBC ≥3.5 x10^9/L
  3. Platelet count ≥ 80x10^9/L
  4. Total bilirubin ≤1.5xULN
  5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 times upper limit of normal (ULN)
  6. BUN≤1.5xULN
  7. Serum creatinine ≤1.5xULN or creatinine clearance ratio ≥60 mL/min
* Any prior treatment (chemotherapy, radiotherapy or surgery) must be completed over 4 weeks(target therapy over 2 weeks) from the screening; Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1 (CTCAE v 4.03)
* International normalized ratio (INR) ≤ 1.5
* Patients and their partners should be willing to use methods of contraception or total abstinence from start of dosing until 6 months after discontinuing of study treatment

Exclusion Criteria:

* Prior treated with AC0010 or allergic to drug or its formulation ingredients
* Patients receiving other anti-tumor therapy
* Impairment of GI disease, renal disorders or liver disease that may significantly alter the absorption and metabolic of AC0010 (e.g., Unable to swallow, liver, kidney or gastrointestinal partial resection, chronic diarrhea and intestinal obstruction)
* HCVAb positive, active hepatitis B (excluding HBV carriers), Hepatitis virus markers positive and receiving anti-virus drugs
* Meningeal metastasis; brain metastasis with whole brain radiotherapy; prior received hormones or mannitol for the brain metastasis
* Previous EGFR-TKI treatment related Interstitial lung disease history
* Known human immunodeficiency virus infection (HIV), other acquired or congenital immunodeficiency disease, or a history of organ transplantation
* Any severe and / or uncontrolled active infections
* Patients receiving concomitant immunosuppressive agents or high-dose corticosteroids
* Any severe and / or uncontrolled medical conditions
* Patients being treated with drugs recognized as being inhibitors or inducers of the liver isoenzyme in the last 4 weeks prior to registration in the current study
* Within 3 days prior to the treatment intaking of pitaya, pomelo, grapefruit, orange, mango and other fruit may affect drug metabolizing enzymes or juice
* Within 2 days prior to the treatment intaking of coffee, tea, cola, chocolate, or other caffeine containing beverages, alcoholic beverages and / or other alcoholic products
* Major surgery, incisional biopsy or traumatic injuries;
* Within 4 weeks prior to the screening patients with bleeding ≥ grade 3, non-healing wound, sever ulcer or bone fracture
* Patients received high dose irradiation treatment or other 14C-labeled drug within 1 year
* Known a history of alcoholism or drug abuse
* Nicotine or urine drug testing was positive
* Participate in any clinical trial within 4 weeks prior to the screening
* Investigator judgment that patient is unsuitable to participate in study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics, Cumalative excretion and Metabolite of 14C-labeled AC0010 | up to 8 Days
  Pharmacokinetics of 14C-labeled AC0010 Radioactivity in whole blood and plasma,Cumulative excretion of 14C-labeled AC0010 radioactivity in feces and urine,Metabolite identification of 14C-labeled AC0010 in plasma, urine and feces

SECONDARY OUTCOMES:
Quantitative analysis of plasma concentrations of unlabeled AC0010 | up to 8 Days
  Quantitative analysis of plasma concentrations of unlabeled AC0010 using a validated LC-MS/MS method
Number of adverse events (AE) experienced by patients | up to 8 Days
  Number of adverse events (AE) experienced by patients to assess safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shao, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Yongqian Shu, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Lihua Bao, Doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China